CLINICAL TRIAL: NCT07404046
Title: Comparison of Bone Ingrowth and Intra-articular Remodeling of Autologous Tendon and Muscle-tendon Semitendinosus Graft After Arthroscopic Anterior Cruciate Ligament Reconstruction Surgery
Brief Title: Comparison of Tendon and Muscle-Tendon Semitendinosus Grafts After ACL Reconstruction
Acronym: CandyStripe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Marin Glavčić, Medical Doctor, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/0719-3
Record Dates: First submitted 2025-12-21; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cruciate Ligament Reconstruction
Keywords: Arthroscopy; Tissue Remodeling; Anterior Cruciate Ligament; Semitendinosus Muscle; Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tendon (Active Comparator): Intervention Name: Tendon-only ST graft Procedure/Surgery: Arthroscopic all-inside ACL reconstruction using an autologous semitendinosus tendon graft without meniscus repair.
  Details:
  Standard tendon graft preparation and fixation Tunnel creation and concomitant lateral tenodesis Anesthesia per protocol Standardized post-op rehab
  Interventions: Procedure: ACL reconstruction
- Tendon + meniscus (Active Comparator): Intervention Name: Tendon-only ST graft + meniscus repair Procedure/Surgery: Arthroscopic all-inside ACL reconstruction using an autologous semitendinosus tendon graft with concurrent meniscus suture.
  Details:
  Standard tendon graft preparation and fixation Tunnel creation and concomitant lateral tenodesis Meniscus repair as needed Anesthesia per protocol Standardized post-op rehab
  Interventions: Procedure: ACL reconstruction
- Muscle tendon (Active Comparator): Intervention Name: Muscle-tendon ST graft Procedure/Surgery: Arthroscopic all-inside ACL reconstruction using an autologous semitendinosus graft preserving muscle fibers, without meniscus repair.
  Details:
  Muscle-tendon graft preparation and fixation Tunnel creation and concomitant lateral tenodesis Anesthesia per protocol Standardized post-op rehab
  Interventions: Procedure: ACL reconstruction
- Muscle tendon + meniscus (Active Comparator): Intervention Name: Muscle-tendon ST graft + meniscus repair Procedure/Surgery: Arthroscopic all-inside ACL reconstruction using an autologous semitendinosus graft preserving muscle fibers, with meniscus repair.
  Details:
  Muscle-tendon graft preparation and fixation Tunnel creation and concomitant lateral tenodesis Meniscus repair technique as needed Anesthesia per protocol Standardized post-op rehab
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — Participants will undergo arthroscopic all-inside anterior cruciate ligament reconstruction using an autologous semitendinosus graft. In the experimental intervention, a muscle-tendon semitendinosus graft is used, with preservation of muscle fibers on the tendon. In the control intervention, a standard tendon-only semitendinosus graft is used. In both groups, graft preparation, tunnel creation, fixation technique, and concomitant lateral tenodesis are identical, and all procedures are performed by the same surgeon following a standardized protocol.

SUMMARY:
Aim: Comparison of tendon to bone ingrowth in bone tunnels and intra-articular remodeling of the graft after anterior cruciate ligament surgery with a muscle-tendon graft and those with a tendon graft. Subjects and methods: It is a single-blind prospective randomized study that would include at least 40 patients with an anterior cruciate ligament rupture. Patients would be randomly divided into two groups of minimally 20 patients each. Patients in the first study group would undergo ACL reconstruction with a muscle-tendon graft, while patients in the control group would be treated with the standard method of ACL reconstruction with a tendon graft.

Expected contribution to the field: The assumption is that the obtained results could enable a better understanding of the contribution of remaining muscle fibers on the tendon in anterior cruciate ligament reconstruction operations to the tendon to bone ingrowth and intra-articular remodeling of the graft of operated patients.

DETAILED DESCRIPTION:
This is a prospective, randomized clinical study conducted at Dubrava University Hospital. At least 40 patients aged 18 to 50 years with clinically and MRI-confirmed anterior cruciate ligament rupture and indication for concomitant lateral tenodesis will be enrolled. Participants will be randomly assigned in a 1:1 ratio to undergo arthroscopic all-inside ACL reconstruction using either a muscle-tendon semitendinosus graft (experimental group) or a standard tendon-only semitendinosus graft (control group). All surgical procedures will be performed by the same surgeon and supplemented with modified Lemaire lateral tenodesis.

Clinical assessments will be performed preoperatively and at 6 weeks, 6 and 12 months postoperatively and will include validated patient-reported outcome measures (EQ-5D and KOOS) and a non-validated Croatian version of the IKDC Subjective Knee Evaluation Form. Knee stability will be assessed 12 months postoperatively using a digital Lachmeter device.

Magnetic resonance imaging of the operated knee will be performed at 6 weeks, 6 and 12 months using a standardized 3T MRI protocol including proton density sequences and T2 mapping. Intra-articular graft remodeling will be assessed using the signal-to-noise quotient method, with standardized regions of interest placed at the proximal, middle, and distal portions of the intra-articular graft and at the posterior cruciate ligament. Tendon-to-bone healing will be evaluated by measuring femoral and tibial tunnel diameters and calculating percentage tunnel widening relative to intraoperative tunnel size.

All participants will follow identical postoperative rehabilitation protocols. MRI analysis will be performed by two experienced musculoskeletal radiologists blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and radiologically confirmed anterior cruciate ligament (ACL) rupture.
* Age between 18 and 50 years.
* Intact posterior cruciate ligament and collateral ligaments.
* Signed informed consent to participate in the study.
* Patients meeting at least one indication for concomitant lateral tenodesis, including: age under 25 years, positive pivot-shift test, presence of Segond fracture, participation in sports with frequent changes of direction and rotational knee loads, or joint hypermobility (Beighton score ≥ 7).

Exclusion Criteria:

* Previous ACL reconstruction of the same knee.
* Inability to use a graft prepared by quadruple folding of the semitendinosus tendon.
* Graft diameter < 7.5 mm.
* MRI-confirmed unsuccessful meniscal healing after repair.
* Acute joint infection or history of joint infection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
SNQ | 6 weeks, 6 and 12 months postoperatively
  To analyze and compare T2 signal-to-noise ratio values on magnetic resonance imaging at 6 weeks, 6 and 12 months postoperatively within and between the two study groups. The SNQ is calculated as the ratio of the graft T2 signal intensity to the signal intensity of a reference tissue on MRI. Higher SNQ values indicate higher graft signal, which corresponds to lower graft maturity/quality.
  Scale: Continuous numerical value (exact values depend on MRI signal calibration).

SECONDARY OUTCOMES:
Bone Tunnel Diameter - Femur | 6 weeks, 6 months, 12 months postoperatively
  Description: The diameter of the femoral bone tunnel measured on MRI at 6 and 12 months postoperatively compared to the intraoperatively drilled diameter.
  Units: Millimeters (mm) Directionality: Higher values indicate tunnel widening
Bone Tunnel Diameter - Tibia | 6 weeks, 6 months, 12 months postoperatively
  Description: The diameter of the tibial bone tunnel measured on MRI at 6 and 12 months postoperatively compared to the intraoperatively drilled diameter.
  Units: Millimeters (mm) Directionality: Higher values indicate tunnel widening.
Knee Stability - Anterior Tibial Translation | 12 months postoperatively
  Description: The anterior-posterior stability of the operated knee measured with the Lachmeter device at 12 months postoperatively.
  Units: Millimeters (mm) of anterior tibial translation Directionality: Higher values indicate greater laxity (worse stability)
KOOS - Pain Subscale | Before surgery, 6 weeks, 6 months, 12 months postoperatively
  Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Pain subscale, assessing knee pain.
  Scale: 0-100 (0 = extreme pain, 100 = no pain; higher scores = better outcome)
KOOS - Symptoms Subscale | Before surgery, 6 weeks, 6 months, 12 months postoperatively
  Description: KOOS - Symptoms subscale, assessing knee symptoms (e.g., swelling, stiffness).
  Scale: 0-100 (0 = severe symptoms, 100 = no symptoms; higher scores = better outcome)
KOOS - Activities of Daily Living (ADL) Subscale | Before surgery, 6 weeks, 6 months, 12 months postoperatively
  Description: KOOS - ADL subscale, assessing functional ability in daily activities.
  Scale: 0-100 (0 = extreme limitation, 100 = no limitation; higher scores = better outcome)
KOOS - Sports/Recreation Subscale | Before surgery, 6 weeks, 6 months, 12 months postoperatively
  Description: KOOS - Sports/Recreation subscale, assessing function during sport or recreational activity.
  Scale: 0-100 (0 = extreme limitation, 100 = no limitation; higher scores = better outcome)
KOOS - Quality of Life (QoL) Subscale | Before surgery, 6 weeks, 6 months, 12 months postoperatively
  Description: KOOS - QoL subscale, assessing knee-related quality of life. Scale: 0-100 (0 = extreme problem, 100 = no problem; higher scores = better outcome)
IKDC-SKF (International Knee Documentation Committee - Subjective Knee Form) | Before surgery, 6 weeks, 6 months, 12 months postoperatively
  Description: Patient-reported measure of knee function, symptoms, and sports activity.
  Scale: 0-100 (0 = worst knee function, 100 = best knee function; higher scores = better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided